CLINICAL TRIAL: NCT05325385
Title: An Estimation of the Incidence of Ventricular Fibrillation (VF) at the Initial Time of Collapse in Out-of-Hospital Cardiac Arrest and the Duration of VF Prior to Its Deterioration to a Non-Shockable Rhythm
Brief Title: Ventricular Fibrillation Following Out-of-hospital Cardiac Arrest
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: Warwick University Clinical Trials Unit (Unknown)
Responsible Party: Sponsor
Other Study IDs: IRAS Project ID: 315145
Record Dates: First submitted 2022-04-05; First posted 2022-04-13 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Cardiac Arrest, Out-Of-Hospital; Ventricular Fibrillation
Keywords: Cardiac arrest; Ventricular fibrillation; Ambulance; Survival
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Ventricular Fibrillation; Heart Arrest

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- OHCA attended by ambulance service: All adults attended by ambulance service where time of collapse and initial rhythm is known.
  Interventions: Other: There are no interventions - this is a database study only

INTERVENTIONS:
Other: There are no interventions - this is a database study only — There are no interventions - this is a database study only

SUMMARY:
The majority of survivors suffering an out-of-hospital cardiac arrest (OHCA) are those who initially present with a shockable rhythm, which is usually ventricular fibrillation (VF). When untreated, VF progresses to asystole over a short period of time so the percentage of those with a survivable rhythm also decreases with time.

There is relatively little data exploring the initial rate of VF and the time course of its subsequent progression to a non-shockable rhythm. An understanding of this data will give a better picture of how potentially survivable rhythms (VF) change with time and guide the response times that are required to ensure arrival before VF deteriorates to asystole.

The Investigators will use the UK OHCA outcomes database to examine the percentage of patients presenting with VF as the initial rhythm according to time since collapse in order to establish the rate at which VF deteriorates to asystole.

DETAILED DESCRIPTION:
Patients suffering an out-of-hospital cardiac arrest (OHCA) present in one of two broad groups; non-shockable or shockable rhythms. The former group comprises asystole or pulseless electrical activity (PEA) and the latter, ventricular fibrillation (VF) or ventricular tachycardia (VT). Recent UK data show that the majority present in a non-shockable rhythm (asystole 50.9%, PEA 22.8%) with only 23% in a shockable rhythm, primarily ventricular fibrillation. (VT represents only a small proportion of shockable rhythms).

Whilst survival from any of these rhythms is poor, the majority of survivors are those who initially present with a shockable rhythm. In a recent pooled analysis of the PARAMEDIC2 and PACA trials, 32.8% of those in shockable rhythms achieved ROSC, compared with 46.0% in shockable rhythms. Of those achieving neurologically intact survival only 0.55% of those in non-shockable rhythms did so, compared with 8.63% in shockable rhythms; a 16-fold difference in survival. Therefore the vast majority of those who survive do so because they present in VF, which is potentially a survivable rhythm.

The initial VF is a relatively short-term arrhythmia. As cellular energy reserves become depleted during the cardiac arrest, the myocyte electrical activity declines resulting in low amplitude VF and eventually a cessation, at which time the rhythm changes to asystole. The proportion of patients presenting in ventricular fibrillation decreases with time and therefore the size of the cohort of patients with a potentially survivable rhythm also decreases with time. Clearly the quicker the rescuer response, the more likely the patient is to still be in VF and the more likely this rhythm can be treated successfully. For every minute without CPR, survival from witnessed ventricular fibrillation (VF) cardiac arrest decreases by 7-10%. Once VF deteriorates to asystole, then survival is unlikely.

Most studies documenting the incidence of VF as the presenting rhythm at OHCA report a cumulative value based on the average of the study's EMS response times. There is relatively little data exploring the initial rate of VF and the time course of its subsequent progression to a non-shockable rhythm. Although earlier studies of OHCA reported high rates of initial VF such as a study from Sweden in 2000, which documented an initial rate of 43%, these high initial rates of VF are consistently not reported in current studies, where the incidence is typically 20-25%, despite improvements in the delivery of bystander CPR which can prolong the VF duration. Although there is contemporary data documenting the overall rates of initial VF at OHCA, no current UK study has examined how the incidence of initial VF changes with time from onset of cardiac arrest (as measured from time from collapse).

An understanding of this data will give a better picture of how potentially survivable rhythms (VF) change with time and guide the response times that are required to ensure arrival before VF deteriorates to asystole.

Additionally, an extrapolation of data into the time window prior to ambulance arrival may allow an estimate of the percentage of patients where VF is the initial rhythm at the time of cardiac arrest onset. Although one study has estimated this as 60-70%, and another as high as 80-90%, these estimates are based on data that does not reflect current estimates of VF incidence. There is also little contemporary data on the rate at which VF progresses to asystole when untreated. Again, historic studies have estimated the rate of VF dissolution into asystole of approximately 2% per minute, but this is not consistent with the current relatively low rates of initial VF, the rapid decline in survival with time, even for VF and possible confounding effect of bystander CPR which is not factored in to most studies.

The Investigators will use five years of data from the UK Warwick University OHCA outcomes database to examine the percentage of patients presenting with VF as the initial rhythm according to time since collapse in order to establish the rate at which VF deteriorates to asystole.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* Out-of-hospital cardiac arrest
* Known time of collapse
* Known initial rhythm documented by ambulance crew

Exclusion Criteria:

* Paediatric cases
* Trauma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients in cardiac arrest attended by ambulance services (England) where data has been submitted to the Warwick University OHCA outcomes database.
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Presenting rhythm | From 01.01.2016 to 31.12.2020
  An estimate of the incidence of VF at the initial time of collapse from a out-of-hospital cardiac arrest.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Southampton, Southampton, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Any request for IPD must directed to the Warwick OHCA outcomes database administrator.

REFERENCES:
- See also: Warwick University OHCA outcomes database — https://warwick.ac.uk/fac/sci/med/research/ctu/trials/ohcao/